CLINICAL TRIAL: NCT04453163
Title: Interest of Improved Recovery After Surgery (IRAS) Management [RAAC in French] in Percutaneous Vertebroplasty
Brief Title: Interest of the Patient Management by Improved Recovery After Surgery in Percutaneous Vertebroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2020-A00600-39
Record Dates: First submitted 2020-06-26; First posted 2020-07-01 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Vertebral Compression
MeSH Terms: interventions — Vertebroplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RAAC program (Experimental): If the patient is under the "RAAC" group, he/she will then be received in consultation by a RAAC specialist nurse, between the anesthesia / radiology consultation and the intervention. This RAAC nurse will explain the procedure and show him/her an information video on vertebroplasty. Information about managing anxiety and pain will also be provided. In addition, the day after the patient leaves the clinic, the RAAC nurse will call him/her to inquire.
  Interventions: Procedure: Vertebroplasty
- Standard management program (Other): If the patient is under the "control" group, he/she will be taken care of according to the standard protocol after a surgery in percutaneous vertebroplasty. The patient will not have a consultation with the specialized nurse.
  Interventions: Procedure: Vertebroplasty

INTERVENTIONS:
Procedure: Vertebroplasty — Patient will undergo a surgery in percutaneous vertebroplasty

SUMMARY:
This research aims to demonstrate the benefits of the RAAC program for patients undergoing cementoplasty, in particular on their level of anxiety and pain control throughout the perioperative phase.

DETAILED DESCRIPTION:
The aim of the study is to compare the preoperative anxiety of patients hospitalized for a percutaneous vertebroplasty, depending on whether or not they are managed in an RAAC program.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 80 years or ≥ 18 years with oncological history;
* Patient with vertebral compression fracture with indication for percutaneous vertebroplasty;
* Patient seen in preoperative anesthesia / radiology consultation more than 4 days before the date of the vertebroplasty;
* Having expressed their consent to participate in the study.

Exclusion Criteria:

* Patient with a contraindication to percutaneous vertebroplasty, such as coagulation disorders, or an allergy or hypersensitivity to any of the products administered during the procedure;
* Patient not affiliated to a social security scheme;
* Patient participating in another clinical trial during the follow-up period;
* Inability to understand information related to the study (linguistic, psychiatric, cognitive reason, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-11-17 (Actual); Primary Completion 2022-12-19 (Actual); Study Completion 2022-12-19 (Actual)

PRIMARY OUTCOMES:
Superiority of Improved Recovery After Surgery versus standard management over preoperative anxiety | 10 days
  The main analysis consists of testing the superiority of Improved Recovery After Surgery versus standard management over preoperative anxiety, evaluated on a numerical scale of 0 to 10

SECONDARY OUTCOMES:
Pain evaluation | 10 days
  Evaluation of the pain on a numerical scale of 0 - no pain to 10 - maximum pain imaginable
Patient satisfaction | 10 days
  Evaluation of the patient satisfaction with care, assessed on a 5-level scale (not at all satisfied / somewhat dissatisfied / moderately satisfied / somewhat satisfied / very satisfied)
Functional impotence | 10 days
  Evaluation of the functional impotence of low back pain by the Quebec score, which includes 20 questions on the ability to undertake daily activities, rated from 0 (no difficulty) to 5 (unable). The score therefore varies from 0 to 100.
Consumption of analgesics | 10 days
  Evaluation of the consumption of analgesics expressed in mg of morphine equivalent.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique Belharra, Bayonne, France

IPD SHARING:
Plan to Share IPD: No